CLINICAL TRIAL: NCT04262973
Title: Interprofessional Education and Collaborative Practice Model for Dementia in Acute Care: Development, Implementation and Evaluation
Brief Title: Interprofessional Education and Collaborative Practice Model for Dementia in Acute Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KMUHIRB-SV(1)-20170070
Record Dates: First submitted 2020-02-04; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Dementia
Keywords: dementia; hospital; acute care; interprofessional education; interprofessional practice
MeSH Terms: conditions — Dementia | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experimental group will not only receive six-hour dementia care course, but also a half-day interprofessional education workshop, maintain a six-month interprofessional practice model, and join interprofessional practice experience-sharing conferences.
  Interventions: Other: education and workshop
- control group (Active Comparator): The control group will only receive six-hour dementia care course.
  Interventions: Other: education

INTERVENTIONS:
Other: education — six-hour dementia care course
  Arms: control group
Other: education and workshop — six-hour dementia care course, half-day interprofessional education workshop, and interprofessional practice
  Arms: experimental group

SUMMARY:
The purpose of this study is to develop an interprofessional education and practice model for acute care related to dementia and evaluate its effectiveness of implementation.

DETAILED DESCRIPTION:
The researchers will recruit participants from a medical center (experimental group) and two regional hospitals (control group) in southern Taiwan. Both the experimental group and the control group will contain 150 healthcare professionals and 64 patients with dementia. Both of the groups will receive a six-hour dementia care course. Then, only the experimental group will receive a half-day interprofessional education workshop, maintain a six-month interprofessional practice model, and join interprofessional practice experience-sharing conferences. The evaluation of outcomes will include the analyses of healthcare professionals' knowledge, attitudes, and self-efficacy of dementia care. The evaluation times are to be before and after the dementia care course and after the six months of interprofessional practice. The other evaluation of outcome is comparison of the outcomes of hospitalized patients with dementia between the two groups before the interprofessional education workshop and after the interprofessional practice.

ELIGIBILITY:
Inclusion Criteria:

* healthcare professionals having worked for 3 months or more
* emergency/hospitalized patients with dementia
* patients diagnosed dementia
* scoring 1 or more in Clinical Dementia Rating (CDR).

Exclusion Criteria:

* healthcare professionals working in obstetrics, pediatrics, outpatient, or hemodialysis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Change of Dementia Care Knowledge | Before education program(pre-intervention), after education program(10 months), after the workshop(10 months), after the six months interprofessional practice(post intervention)[about 8 months]
  testing the change of professionals' Dementia Care Knowledge. The minimum value of this scale is 0, and the maximum value is 16.
  Higher scores mean having better Dementia Care Knowledge.

SECONDARY OUTCOMES:
Change of dementia self-efficacy scale | Before education program(pre-intervention), after education program(10 months), after the workshop(10 months), after the six months interprofessional practice(post intervention)[about 8 months]
  testing professionals' dementia self-efficacy. The scale has not developed yet. It will be developed and test the reliability and validity in this study.
mortality rate of hospitalized patients with dementia | about 2 years
  understand the treatment outcomes of hospitalized patients with dementia before the interventions six months and after interventions six months.
length of stays of hospitalized patients with dementia | about 2 years
  understand the treatment outcomes of hospitalized patients with dementia before the interventions six months and after interventions six months.
the incidence of fall hospitalized patients with dementia | about 2 years
  understand the treatment outcomes of hospitalized patients with dementia before the interventions six months and after interventions six months.
the incidence of pain hospitalized patients with dementia | about 2 years
  understand the treatment outcomes of hospitalized patients with dementia before the interventions six months and after interventions six months.
score of Beck depression inventory | about 2 years
  testing psychological symptoms of hospitalized patients with dementia
score of Cohen-Mansfield Agitation Inventory (CMAI) | about 2 years
  testing behavioral symptoms of hospitalized patients with dementia

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan